CLINICAL TRIAL: NCT01264458
Title: Microvesicle Production After Acute Trauma and Its Clinical Impact on Venothromboembolism
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Myung S. Park, Assistant Professor of Surgery, Mayo Clinic
Other Study IDs: 10-001889
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Venothromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traumatic Injury: Trauma patients arriving at Saint Mary's Emergency Department
- Control group

SUMMARY:
The purpose of this research study is to look at how trauma affects the ability of blood to clot. The blood of people who suffer a traumatic injury can under-clot or over-clot, and this research study will look at blood drawn from people after they suffer a traumatic injury to see how well their blood clots.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years of age or older
* Blunt trauma patients including those with closed head injury
* Penetrating trauma patients

Exclusion Criteria:

* Are on therapeutic anticoagulation
* Have preexisting coagulopathy
* Patients greater than 12 hours from time of injury
* Have history of malignancy or preexisting diagnosis of sepsis or renal failure
* Patients with burn injuries
* Male and female patients younger than 18 years of age
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Trauma patients arriving to Saint Mary's Emergency Department and control patients.
Sampling Method: Probability Sample
Enrollment: 1234 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12-14 (Actual); Study Completion 2014-12-14 (Actual)

PRIMARY OUTCOMES:
Estimate the distribution over time of procoagulant Microvesicles (MVs) concentration by cell of origin and endogenous thrombin potential (ETP). | 6 months
Determine the cumulative incidence of Venothromboembolism (VTE) within three months after major trauma and test the distribution of procoagulant MV concentration and endogenous thrombin generation potential over time as potential predictors of VTE. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Myung Park, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials